CLINICAL TRIAL: NCT06612658
Title: A Prospective, Randomized Double-Blind, Placebo-Controlled, Cross-Over Study to Evaluate Acute Effect of Capsimax on Resistance Exercise Performance, Muscle Oxygenation, Nitric Oxide Release, Resting Energy Expenditure and Reaction Time
Brief Title: Acute Effect of Capsimax on Resistance Exercise Performance, Muscle Oxygenation, Nitric Oxide Release, Resting Energy Expenditure and Reaction Time
Acronym: Capsimax
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hofstra University (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Adam Gonzalez, Associate Professor, Hofstra University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 20240805-AHK-SHS-GON-1; HO-01 (Other Grant/Funding Number: OmniActive Health Technologies)
Record Dates: First submitted 2024-09-10; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: None Volunteer
Keywords: capsaicin; capsimax
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capsimax (Experimental): Capsules containing either 100 mg Capsimax (OmniActive Health Technologies)
  Interventions: Dietary Supplement: A novel, proprietary encapsulated form of Capsicum extract in beadlet form standardized to 2% capsaicinoids
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: A novel, proprietary encapsulated form of Capsicum extract in beadlet form standardized to 2% capsaicinoids

INTERVENTIONS:
Dietary Supplement: A novel, proprietary encapsulated form of Capsicum extract in beadlet form standardized to 2% capsaicinoids — This study will investigate the effect of the supplement on exercise performance.
  Other Names: Capsimax; Capsaicin

SUMMARY:
Capsimax is a novel, proprietary encapsulated form of capsaicin, a natural and bioactive phytochemical found in chili pepper and other spicy food. The purpose of this study is to investigate the effect of Capsimax on resistance exercise performance, reaction time, and resting energy expenditure around exercise. This investigation will also measure muscle oxygenation and intramuscular nitric oxide in real time during resistance exercise using a non-invasive wearable technology.

Primary Objective • To examine the effects of Capsimax on physical performance metrics including peak power and rate of force development during an isometric strength test and performance during the barbell back squat exercise protocol (e.g., repetitions performed, total volume, peak power, average power).

Secondary Objectives

* To examine the effects of Capsimax on resting energy expenditure around exercise.
* To examine the effects of Capsimax on nitric oxide bioavailability and skeletal muscle oxygenation during exercise.

Exploratory Objective

• To examine the effects of Capsimax on reaction time around exercise

DETAILED DESCRIPTION:
Capsimax is a novel, proprietary encapsulated form of capsaicin, a natural and bioactive phytochemical found in chili pepper and other spicy food. The purpose of this study is to investigate the effect of Capsimax on resistance exercise performance, reaction time, and resting energy expenditure around exercise. This investigation will also measure muscle oxygenation and intramuscular nitric oxide in real time during resistance exercise using a non-invasive wearable technology.

Primary Objective • To examine the effects of Capsimax on physical performance metrics including peak power and rate of force development during an isometric strength test and performance during the barbell back squat exercise protocol (e.g., repetitions performed, total volume, peak power, average power).

Secondary Objectives

* To examine the effects of Capsimax on resting energy expenditure around exercise.
* To examine the effects of Capsimax on nitric oxide bioavailability and skeletal muscle oxygenation during exercise.

Exploratory Objective

• To examine the effects of Capsimax on reaction time around exercise

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged between 18-35 years (both limits inclusive).
2. Subjects must have a BMI of 18.5 to 29.9 kg/m2 (both limits inclusive)
3. Subjects must have greater than one year of resistance training experience at a frequency of 2 days per week.
4. Subjects must be proficient in the barbell back squat exercise.
5. Subjects must be free of any physical limitations or chronic illness that may affect performance.
6. Subjects must be free of any medications.
7. Subjects who agree to refrain from consuming alcohol 24 hours prior to the visit days.
8. Subjects who agreed to refrain from consuming caffeine and caffeine-containing products 12 hour prior to visit days
9. Subject willing to provide written consent.

Exclusion Criteria:

1. Subjects who have hypersensitivity or history of allergy to the study product.
2. Subjects with inability to swallow soft gel capsules.
3. Subjects with any other medical condition that might adversely impact the safety of the study participants or confound the study results.
4. Subjects who require medications.
5. Subjects who regularly use a dietary supplement containing Capsimax or other ingredients that would impact study endpoints.
6. Subjects who had been treated with any investigational drug or investigational device within a period of 3 months prior to study entry

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Resistance exercise performance | 1 day
  Performance during the barbell back squat exercise protocol (e.g., repetitions performed, total volume, peak power, average power).
Isometric strength test | 1 day
  Physical performance metrics will be assessed during an isometric mid-thigh pull test including peak power and rate of force development

SECONDARY OUTCOMES:
Energy expenditure | 1 day
  Resting energy expenditure metrics
Nitric oxide release and skeletal muscle oxygenation | 1 day
  Prior to initiating the barbell back squat exercise protocol, participants will have a sensor (NNOXX One, NNOXX Inc.) secured to a standardized position on the thigh to measure nitric oxide release and muscle oxygenation (i.e., a measure of how much blood and oxygen is being delivered to the working muscle) during exercise. This is a non-invasive device that adheres to the skin with tape and allows for real-time feedback regarding the status of the muscle (Figure 1). NNOXX One utilizes spectrometer and optical sensors to non-invasively measure muscle oxygenation and nitric oxide by analyzing the absorption and reflection of light interacting with bodily tissues.
Subjective feelings of pain and rating of perceived exertion | 1 day
  Questionnaires will be provided prior to supplementation, prior to exercise, and following the resistance exercise protocol. Participants will be instructed to assess their subjective feelings of fatigue and pain using a 15-cm visual analog scale (VAS). The scale will be anchored by the words "low" and "high" to represent extreme ratings where the greater measured value represents a greater feeling. Questions will be structured as "My level of fatigue is." Participants will be asked to rate their feelings at each time point by marking on the corresponding line. A rating of perceived exertion (RPE) will also be recorded following the resistance exercise protocol.

OTHER OUTCOMES:
Reaction time | 1 day
  Reaction time will be assessed with a visual-cognitive reactionary test

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Gonzalez, PhD, Principal Investigator — Hofstra University
Locations (1):
- Hofstra University, Hempstead, New York, United States

IPD SHARING:
Plan to Share IPD: No